CLINICAL TRIAL: NCT03421938
Title: Investigation of the Effect of Downhill-uphill Walking Exercises on Functional Level and Muscle Strength in Patients With Knee Arthroplasty.
Brief Title: Effect of Downhill-uphill Walking Exercises on Functional Level and Muscle Strength in Patients With Knee Arthroplasty.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: I changed my PhD thesis
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Abdurrahman Nalbant, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3243-GOA
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Knee Arthroplasty
Keywords: total knee arthroplasty; walking exercises; uphill-downhill walking exercises; functional level

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Downhill Exercise Group) (Experimental): This group will have downhill walking exercises with %10 slope.
  Interventions: Other: Walking Exercise
- Group 2 ( Uphill Exercise Group) (Experimental): This group will have uphill walking exercises on the treadmill with %10 slope.
  Interventions: Other: Walking Exercise

INTERVENTIONS:
Other: Walking Exercise — Group 1 will have downhill walking exercises with %10 slope; group 2 uphill walking exercises on the treadmill with %10 slope..

SUMMARY:
This study is planned for investigating effect of downhill-uphill walking exercises on functional level and muscle strength in patients with knee arthroplasty. Patients who have had primary knee arthroplasty and has gone 3 months after surgery will be included in this study. The patients will be divided into two groups by randomization. Totally, 22 patients will be included in this study. Every patients will have same standart post-operative rehabilitation programme. In addition,group 1 will have downhill walking exercises with %10 slope; group 2 uphill walking exercises on the treadmill with %10 slope. Assessments will be made before and after treatment.

DETAILED DESCRIPTION:
This study is planned for investigating effect of downhill-uphill walking exercises on functional level and muscle strength in patients with knee arthroplasty. Patients who have had primary knee arthroplasty and has gone 3 months after surgery will be included in this study. The patients will be divided into two groups by randomization. Totally, 22 patients will be included in this study. Every patients will have same standart post-operative rehabilitation programme. Assessments will be made before and after treatment. Rehabilitation programme after knee arthroplasty has included muscle strength and endurance, balance and proprioceptive sensation, increasing functional level and providing independence in daily life activities.For this purpose, a standard physiotherapy program will be implemented in accordance with the goals and objectives stated for all patients. In addition,group 1 will have downhill walking exercises with %10 slope; group 2 uphill walking exercises on the treadmill with %10 slope. It takes 30 minutes for one session.

Exercise intensity was measured before treatment; will be determined using the Karvonen formula depending on the heart rate. Walking intensity during exercise; 55% of the maximum heart rate will be determined at the beginning of the treatment and 85% towards the end of the treatment. Walking exercise on the treadmill will be performed in conjunction with a qualified physiotherapist in this area for 4 weeks(3 session in 1 week).

Within the scope of the assessments, patients' pain levels will be determined using the Numeric Pain Scale (NAS). For the knee joint, the normal range of motion will be determined by universal goniometer. For the determination of functional level, Iowa functional activity scale, Iowa ambulatory speed scale and Hospital For Special Surgery (HSS) knee scoring, 10-meter walking speed, Timed Up and Go (TUG) test, SF-12(12-Item Short Form Survey) quality of life scale will be used. Hand dynamometer will be used to evaluate muscle strength.These assessments will be made before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative diagnosis have to be knee osteoarthritis.
* Patients with primary knee arthroplasty after 3 months surgery.

Exclusion Criteria:

* BMI >40 kg/m2
* Having orthopedic or neurologic disorders which cause walking disorders.
* Revision total knee arthroplasty

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-03-20 (Estimated); Study Completion 2018-03-20 (Estimated)

PRIMARY OUTCOMES:
Change of Iowa Level of Assistance Scale | Change from Baseline Patient's Functional Level at 4 weeks
  This test assesses the patient's ability to perform four functional activities, namely, supine to sitting on the edge of the bed,sitting on the edge of the bed to standing, walking 4.57 metres. The scoring of these activities is done as independent 6 points, observational aid 5 points, minimum help 4 points, medium help 3 points, maximum help 2 points, fail 1 point and untest 0 points. Higher values represent a better outcome.
  Speed scoring is done by evaluating the walking speed at a distance of 13.4 meters (44 steps). 20 seconds (sec) and below are recorded as 0, 21-30 sec 1, 31-40 sec 2, 41-50 3, 51-60 sec 4, 61-70 sec 5 and 70 sec. Higher values represent a worse outcome
Change of Hospital For Special Surgery Knee Score | Change from Baseline Patient's Functional Level at 4 weeks
  Hospital for Special Surgery knee score. A scoring system evaluation of pain, mobility, range of motion and deforming of the knee giving 0-100 points
Change of 10 meter walk speed test | Change from Baseline Patient's Functional Level at 4 weeks
  Individual walks without assistance 10 meters and the time is measured for the intermediate 6 meters to allow for acceleration and deceleration, start timing when the toes of the leading foot crosses the 2-meter mark, stop timing when the toes of the leading foot crosses the 8-meter mark,assistive devices can be used but should be kept consistent and documented from test to test, if physical assistance is required to walk, this should not be performed can be performed at preferred walking speed or fastest speed possible documentation should include the speed tested (preferred vs. fast) collect three trials and calculate the average of the three trials
Change of Timed Up and Go (TUG) | Change from Baseline Patient's Functional Level at 4 weeks
  To determine fall risk and measure the progress of balance, sit to stand, and walking.The patient starts in a seated position. The patient stands up upon therapist's command walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. The subject is allowed to use an assistive device.

SECONDARY OUTCOMES:
SF-12 | Change from Baseline SF-12 score Level at 4 weeks
  SF-12 Health Survey is a shorter version of the SF-36 Health Survey that uses just 12 questions to measure functional health and well-being from the patient's point of view. The SF-12 is a practical, reliable and valid measure of physical and mental health and is particularly useful in large population health surveys or for applications that combine a generic and disease-specific health survey.
Numeric Pain Scale | Change from Baseline Patient's Pain Level at 4 weeks
  Severity of pain was rated by each patient marking their current level of pain on a 10cm visual analogue scale (VAS), where 0 represented no pain and 10 was the worst pain imaginable.Higher values represent a worse outcome.
Range of Motion | Change from Baseline Patient's Range of Motion 4th week
  Each patient's active (unassisted) range of knee extension and flexion will be measured, using a goniometer with the patient in the supine position.
Muscle Strength | Change from Baseline Patient's Muscles Strengths at 4 weeks
  Strength of knee muscles will be evaluated by hand-held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahman Nalbant, PT,MSc, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Shields RK, Enloe LJ, Leo KC. Health related quality of life in patients with total hip or knee replacement. Arch Phys Med Rehabil. 1999 May;80(5):572-9. doi: 10.1016/s0003-9993(99)90202-2. PMID 10326924
- [Background] Moffet H, Collet JP, Shapiro SH, Paradis G, Marquis F, Roy L. Effectiveness of intensive rehabilitation on functional ability and quality of life after first total knee arthroplasty: A single-blind randomized controlled trial. Arch Phys Med Rehabil. 2004 Apr;85(4):546-56. doi: 10.1016/j.apmr.2003.08.080. PMID 15083429
- [Background] Noble PC, Gordon MJ, Weiss JM, Reddix RN, Conditt MA, Mathis KB. Does total knee replacement restore normal knee function? Clin Orthop Relat Res. 2005 Feb;(431):157-65. doi: 10.1097/01.blo.0000150130.03519.fb. PMID 15685070
- [Background] Wylde V, Dieppe P, Hewlett S, Learmonth ID. Total knee replacement: is it really an effective procedure for all? Knee. 2007 Dec;14(6):417-23. doi: 10.1016/j.knee.2007.06.001. Epub 2007 Jun 26. PMID 17596949
- [Background] Petterson SC, Mizner RL, Stevens JE, Raisis L, Bodenstab A, Newcomb W, Snyder-Mackler L. Improved function from progressive strengthening interventions after total knee arthroplasty: a randomized clinical trial with an imbedded prospective cohort. Arthritis Rheum. 2009 Feb 15;61(2):174-83. doi: 10.1002/art.24167. PMID 19177542
- [Background] Yoshida Y, Mizner RL, Ramsey DK, Snyder-Mackler L. Examining outcomes from total knee arthroplasty and the relationship between quadriceps strength and knee function over time. Clin Biomech (Bristol). 2008 Mar;23(3):320-8. doi: 10.1016/j.clinbiomech.2007.10.008. Epub 2007 Dec 3. PMID 18060669
- [Background] Rossi MD, Hasson S. Lower-limb force production in individuals after unilateral total knee arthroplasty. Arch Phys Med Rehabil. 2004 Aug;85(8):1279-84. doi: 10.1016/j.apmr.2003.11.034. PMID 15295753
- [Background] Mizner RL, Petterson SC, Snyder-Mackler L. Quadriceps strength and the time course of functional recovery after total knee arthroplasty. J Orthop Sports Phys Ther. 2005 Jul;35(7):424-36. doi: 10.2519/jospt.2005.35.7.424. PMID 16108583
- [Background] Meier WA, Marcus RL, Dibble LE, Foreman KB, Peters CL, Mizner RL, LaStayo PC. The long-term contribution of muscle activation and muscle size to quadriceps weakness following total knee arthroplasty. J Geriatr Phys Ther. 2009;32(2):79-82. PMID 20039587
- [Background] Berth A, Urbach D, Awiszus F. Improvement of voluntary quadriceps muscle activation after total knee arthroplasty. Arch Phys Med Rehabil. 2002 Oct;83(10):1432-6. doi: 10.1053/apmr.2002.34829. PMID 12370881
- [Background] Mizner RL, Petterson SC, Stevens JE, Axe MJ, Snyder-Mackler L. Preoperative quadriceps strength predicts functional ability one year after total knee arthroplasty. J Rheumatol. 2005 Aug;32(8):1533-9. PMID 16078331
- [Background] LaStayo P, Marcus R, Dibble L, Frajacomo F, Lindstedt S. Eccentric exercise in rehabilitation: safety, feasibility, and application. J Appl Physiol (1985). 2014 Jun 1;116(11):1426-34. doi: 10.1152/japplphysiol.00008.2013. Epub 2013 Jul 3. PMID 23823152
- [Background] Rodio A, Fattorini L. Downhill walking to improve lower limb strength in healthy young adults. Eur J Sport Sci. 2014;14(8):806-12. doi: 10.1080/17461391.2014.908958. Epub 2014 Apr 23. PMID 24754630
- [Background] Samaei A, Bakhtiary AH, Hajihasani A, Fatemi E, Motaharinezhad F. Uphill and Downhill Walking in Multiple Sclerosis: A Randomized Controlled Trial. Int J MS Care. 2016 Jan-Feb;18(1):34-41. doi: 10.7224/1537-2073.2014-072. PMID 26917996
- [Background] Langhammer B, Stanghelle JK. Exercise on a treadmill or walking outdoors? A randomized controlled trial comparing effectiveness of two walking exercise programmes late after stroke. Clin Rehabil. 2010 Jan;24(1):46-54. doi: 10.1177/0269215509343328. Epub 2009 Dec 21. PMID 20026572
- [Background] Wiik AV, Aqil A, Tankard S, Amis AA, Cobb JP. Downhill walking gait pattern discriminates between types of knee arthroplasty: improved physiological knee functionality in UKA versus TKA. Knee Surg Sports Traumatol Arthrosc. 2015 Jun;23(6):1748-55. doi: 10.1007/s00167-014-3240-x. Epub 2014 Aug 27. PMID 25160471